CLINICAL TRIAL: NCT06919952
Title: A Cluster-randomized Control Trial of a Workplace Resilience Intervention for Child Care Providers' Mental Health & Well-being
Brief Title: Comparing a Workplace Resilience and a Physical Activity Intervention on Early Childhood Educators Well-being
Acronym: OnWARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 25-0016; R01AT012620 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Resilience
Keywords: child care provider well-being; child care centers; early childhood education; physical activity; resilience; behavior change
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience (Experimental): Centers randomized to Resilience will receive the Stress Management And Resilience Training program. Participating staff will be led through the program by a behavioral health counselor for 3 months. This counselor will orient participants to the Resilience program and the 4 modules. The counselor will also provide 4 coaching calls with directors (at the start of each module). Additionally, the counselor will provide a webinar every 3 weeks (at the end of each module) to all participants. Participants will have access to video lessons and resources. They will receive weekly reminders and encouragement through text messages.
  Interventions: Behavioral: Resilience
- Physical Activity (Active Comparator): Centers randomized to the control arm will receive a physical activity program. Participating staff will be led through the program by a behavioral health counselor for 3 months. This counselor will orient participants to the physical activity program and the 4 modules. The counselor will also provide 4 coaching calls with directors (at the start of each module). Additionally, the counselor will provide a webinar every 3 weeks (at the end of each module) to all participants. Participants will have access to video lessons and resources. They will receive weekly reminders and encouragement through text messages.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Resilience — The Resilience program focuses on drawing on resilience assets and resources, both internal and external. Participants will have access to materials (e.g., lessons, videos, webinars, coaching calls) supporting the adoption of strategies for improving well-being. Behavior change strategies used are meant to increase intervention adherence and improve well-being and resilience.
  Arms: Resilience
Behavioral: Physical Activity — The Physical Activity program focuses on supporting physical activity health habits. Participants will have access to materials (e.g., lessons, videos, webinars, coaching calls) supporting the adoption of strategies of evidence-based strategies for physical activity goals. Behavior change strategies used are meant to help establish, improve or maintain healthy physical activity habits.
  Arms: Physical Activity

SUMMARY:
The goal of this 15-month cluster clinical trial is to compare a resilience and stress management program to a physical activity program for early childhood education (ECE) staff on change in well-being. It will also look to see if changes in well-being continue over time.

The study sample will include 80 child care centers. Including 80 ECE center directors and approximately 560 ECE center staff.

Some ECE centers will receive only the remotely delivered Resilience program. This program works with ECE staff and helps them recognize and strengthen their resilience assets and resources. Other ECE centers will receive only the remotely delivered Physical Activity program that will focus on staff physical activity habits and strength training.

There will be 3 months of active program participation and 12 months of a maintenance period where participants will only have access to program materials.

DETAILED DESCRIPTION:
This study is two-group clustered randomized trial comparing two remotely delivered programs to early childhood education (ECE) center staff, a Resilience program and a Physical Activity program, on ECE center staff change in well-being. The investigators will randomized (by center 1:1 ratio) 80 ECE centers, including 640 ECE staff from these centers, to one of arms (Resilience or Physical Activity) for a 15 month trial (3 months active intervention and 12 months maintenance period). The specific aims are to 1) increase resilience assets and resources for ECE staff, 2) increase overall well-being and organizational assets and resources, and 3) maintain increases in resilience assets and resources, well-being, and organizational assets and resources for ECE staff over time.

Once randomized, all program tasks and activities will be remotely delivered, and guidance will be provided by a behavioral health counselor. Participants will complete their assigned program over four modules spanning 3 months (3 weeks per module). Activities will include an orientation, modules consisting of video lessons and resources, 3 webinars for all participants, text messages (3-5 per week), and 4 coaching calls for ECE center directors only.

Measures will be collected at four timepoints: baseline (0 months), post-intervention (3 months), and long-term maintenance (9 and 15 months). Secondary outcomes will include changes in overall mental health, negative and positive mental health indicators, social support, and organizational assets and resources. Additionally, potential moderators' (e.g., sociodemographic, social determinants of health) influence on treatment effects will be explored. The Reach Effectiveness-Adoption Implementation Maintenance (RE-AIM) Framework will be used to determine reach and representativeness, and potential for organizational level adoption, implementation, and maintenance of the SMART program.

Primary analyses will involve testing change in the total score from the Connor- Davidson Resilience Scale (CD-RISC) between Resilience and Physical Activity arms at 3 months. Using maximum likelihood methods, multi-level linear mixed models (PROC MIXED) that include random effect for cluster to account for covariance between participants within the same center as well as fixed effects for time (0, 3, 9, 15 months), trial arm (resilience or physical activity), time*arm interaction will be used. Similar analyses will be completed for secondary outcomes. Baseline variables including center and worker demographics and social determinants of health will be included as covariates to assess their potential moderating effect.

ELIGIBILITY:
Inclusion Criteria:

Child Care Centers

* Licensed with no plans to close in the next 2 years
* Been in operation for at least 1 year
* Has at least 4 employees

ECE Staff

* Must be at least 18 years old
* Be able to read and speak English
* Must have access to an online resource (e.g., smartphone, tablet, computer)
* Must be willing to receive text messages

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change in Resilience from Baseline to 3 months | Baseline and 3 months
  Resilience of ECE staff will be assessed using the Connor-Davidson Resilience Scale (CD-RISC). ECE staff will fill out through an online survey. The CD-RISC is a 25-item scale. Scores range from 0-100 with higher scores reflecting greater resilience.

SECONDARY OUTCOMES:
Change in Resilience from 3 months to 9 months | 3 months and 9 months
  Resilience of ECE staff will be assessed using the Connor-Davidson Resilience Scale (CD-RISC). ECE staff will fill out through an online survey. The CD-RISC is a 25-item scale. Scores range from 0-100 with higher scores reflecting greater resilience.
Change in Resilience from 9 to 15 months | 9 months and 15 months
  Resilience of ECE staff will be assessed using the Connor-Davidson Resilience Scale (CD-RISC). ECE staff will fill out through an online survey. The CD-RISC is a 25-item scale. Scores range from 0-100 with higher scores reflecting greater resilience.
Change in Well-Being from Baseline to 3 months | Baseline and 3 months
  Global assessment of well-being will be measured through the General Health Questionnaire. This is a 30-item survey captures a broad spectrum of psychological distress encompassing emotional, cognitive, and social aspects of mental health. Scores range from 0-90, with higher scores indicating greater psychological distress.
Change in Organizational Support and Resources from Baseline to 3 months | Baseline and 3 months
  Organizational support and resources will be assessed using the NIOSH worker well-being questionnaire (WellBQ). Specifically, eight Likert-type items from the supportive work culture and health culture at work sections of the survey will be averaged to create this outcome. Items are rated on 1 to 4 scale from strongly disagree to strongly agree, with the final outcome being an average score ranging from 1.00 to 4.00.
Absenteeism from Baseline to 3 months | Baseline to 3 months
  Staff absenteeism will be assessed by asking staff how often they "missed a full day of work" and "missed 1/2 day of work" in the past 4 weeks. Directors will also be asked "On average, how many days per month do staff miss a full day of work when scheduled to be at your center?". Items will be combined to estimate "Days per month staff missed work" at a center.
Staff Turnover rate from Baseline to 3 months | Baseline to 3 months
  Staff turnover will be assessed by asking directors: "How many total staff work at center?" "How many staff have left, quit, or been fired in the past 3 months?", and "how many of those staff have you replaced in the past three months or are currently trying to replace?". Questions will be asked at baseline and 3 month follow-up. Turnover rate for a center will be expressed as: ((# staff left job-(#staff not need replacing)/(# total staff)) * 100 = % turnover.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Hales, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Deborah Jones, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center for Health Promotion and Disease Prevention, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina-Chapel Hill (UNC-CH).
Supporting Information: Study Protocol
Time Frame: Beginning at 9 months and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC-CH.